CLINICAL TRIAL: NCT02109016
Title: A Single Arm, Open-label, Phase 2 Study to Assess the Efficacy and Safety of Lucitanib Given Orally as a Single Agent to Patients With Advanced/Metastatic Lung Cancer and FGF, VEGF, or PDGF Related Genetic Alterations
Brief Title: A Study to Assess the Efficacy and Safety of the VEGFR-FGFR Inhibitor, Lucitanib, Given to Patients With Advanced/Metastatic Lung Cancer and FGF, VEGF, or PDGF Related Genetic Alterations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-3810-II-02
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Non-Small Cell Lung Cancer; Squamous Non-Small Cell Lung Cancer; NSCLC; Small Cell Lung Cancer; SCLC; Lung Cancer; Advanced Lung Cancer; Metastatic Lung Cancer; Stage IV Lung Cancer
Keywords: FGFR1 amplification; FGF alteration; VEGF alteration; PDGF alteration; Tyrosine kinase inhibitor; VEGFR inhibitor; FGFR inhibitor; PDGFR inhibitor; VEGFR-FGFR inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms | interventions — E-3810

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lucitanib (Experimental): Lucitanib given orally once daily on a continuous schedule. Starting dose is 10 mg/day.
  Interventions: Drug: Lucitanib

INTERVENTIONS:
Drug: Lucitanib — Lucitanib given orally to all patients, once daily (q.d.), on a continuous schedule over 28-day cycles, in fasting conditions (at least 2 hours prior to and 2 hours after any meal), until progressive disease or unacceptable toxicity.
  Starting dose is 10 mg/day and can be reduced in 2.5 mg decrements to 5 mg/day based on individual tolerability.

SUMMARY:
The purpose of this study is to determine whether lucitanib is safe and effective in the treatment of patients with advanced/metastatic lung cancer and fibroblast growth factor (FGF), vascular endothelial growth factor receptor (VEGF), or platelet derived growth factor (PDGF) related genetic alterations.

DETAILED DESCRIPTION:
Lucitanib is an oral inhibitor of the tyrosine kinase activity of FGFR 1-3, VEGFR 1-3, and PDGFR α/β. Lucitanib has demonstrated potent anti-tumor and anti-angiogenic activity in vitro proliferation assays and in vivo using human tumor xenograft models, with a trend for stronger efficacy in those with genomic aberrancies of FGF or PDGF. Abnormalities in the FGF, VEGF, and PDGF-related genes are observed across lung cancer histologies.

The first in human trial of lucitanib demonstrated that daily lucitanib is clinically active in patients with advanced solid tumors. Specifically, patients with FGFR1-amplification appeared to derive particular benefit from lucitanib.

Based on these results, this study is designed to explore the safety and anti-tumor activity of daily lucitanib in lung cancer patients with FGF, VEGF, and PDGF genetic alterations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced/metastatic SCLC or NSCLC
* Any of the following tumor tissue based genetic alterations: FGFR1, FGFR2, FGFR3, VEGFA, or PDGFRα amplification; Any FGFR1, FGFR2, or FGFR3 gene fusion; FGFR1, FGFR2, or FGFR3 activating mutation
* Availability of tumor tissue sample suitable for the central confirmation of the genetic alteration and exploratory analyses
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* Measurable disease per RECIST 1.1
* Documented radiographic disease progression following at least one line of therapy in the advanced/metastatic setting

Exclusion Criteria:

* Tumors that are invading a major vessel; NSCLC tumors abutting to a major vessel
* Uncontrolled hypertension, defined as SBP ≥ 140 mmHg and/or DBP ≥ 90 mmHg with optimized anti-hypertensive therapy
* Uncontrolled hypothyroidism defined as serum thyroid stimulating hormone (TSH) higher than 5 mIU/mL while receiving appropriate thyroid hormone therapy
* Symptomatic and/or untreated central nervous system metastases
* Presence of another active cancer
* Ongoing adverse events from surgery or prior anti-cancer therapies, including radiation, targeted, or cytotoxic therapies
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Screening, every 8 weeks; up to 2 years
  Proportion of patients in whom a confirmed Complete Response (CR) or a confirmed Partial Response (PR), as best overall response according to RECIST criteria, is observed.

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Screening, every 8 weeks; up to 2 years
  Proportion of patients in whom a confirmed CR or confirmed PR or a prolonged Stable Disease (SD) (≥ 6 months), as best overall response according to RECIST, is observed
Progression-Free Survival (PFS) | Screening, every 8 weeks; up to 2 years
  Time from the date of first drug intake until the date of progression or death for any cause
Duration of response (DOR) | Screening, every 8 weeks; up to 2 years
  For responders (i.e. patients with best overall response CR or PR), the interval from the time of first documentation of response to the date of progression or death for any cause
Duration of clinical benefit | Screening, every 8 weeks; up to 2 years
  For responders and patients with SD as best overall response, time from the first drug intake until the date of progression or death for any cause
Overall Survival (OS) | Continuously; up to 2 years
  From the date of first drug intake to the date of death for any cause
Tumor growth kinetics | Screening, every 8 weeks; up to 2 years
  Will be evaluated using the following criteria: tumor size; tumor volume; tumor growth
Incidence of adverse events (AEs), clinical laboratory abnormalities, and dose modifications | Continuously; up to 2 years
PK parameters of lucitanib | Cycle 1 Day 14 and 28, Cycle 2 Day 28, Cycle 3 Day 28
Pharmacogenomic analysis of inter-patients variation in gene encoding ADME involved proteins | Cycle 1 Day 1
Pharmacodynamic (PD) evaluation of lucitanib profile | Cycle 1 Day 1 and 14, End of Study
  Soluble growth factors and other biomarkers, including circulating tumor DNA

CONTACTS AND LOCATIONS:
Locations (19):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Associates in Oncology and Hematology, Rockville, Maryland
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
- France (4):
  - CHU Caen, Hôpital de la Côte de Nacre, Caen
  - CHRU Lille, Hôpital Albert Calmette, Lille
  - Hôpital Nord, Marseille
  - Institut Gustave-Roussy, Villejuif
- Germany (3):
  - Universität Duisburg-Essen, Essen
  - Hospital Grosshansdorf, Großhansdorf
  - Pius Hospital Oldenburg, Oldenburg
- Italy (4):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - AOU San Luigi Gonzaga, Orbassano
  - Ospedale S. Maria della Misericordia, Perugia
- Hospital Universitari Vall d'Hebrón, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Liao M, Zhou J, Wride K, Lepley D, Cameron T, Sale M, Xiao J. Population Pharmacokinetic Modeling of Lucitanib in Patients with Advanced Cancer. Eur J Drug Metab Pharmacokinet. 2022 Sep;47(5):711-723. doi: 10.1007/s13318-022-00773-w. Epub 2022 Jul 18. PMID 35844029